CLINICAL TRIAL: NCT02330432
Title: Phase IIb Randomized, Double Blind, Two Arm, Controlled Clinical Trial of Mycobacterium W in Combination With Standard Therapy Versus Standard Therapy Alone in Sepsis
Brief Title: Mycobacterium w in Patients With Severe Sepsis
Acronym: MISS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Collaborators: Pandit Bhagwat Dayal Sharma, PGIMS, Rohtak (Other); St.John's National Academy of Health Sciences (Other)
Responsible Party: Principal Investigator, Ritesh Agarwal, Additional Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pulm/Mw/002
Record Dates: First submitted 2014-12-26; First posted 2015-01-05 (Estimated); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Mycobacterium w vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mycobacterium w group (Experimental): Patients in the experimental arm (Mw) in addition to standard care will receive single daily dose of 0.3 mL of Mw (heat-inactivated Mw [0.5 × 10^9]; Cadila Pharma, Ahmedabad, India) in the deltoid region for 3 consecutive days
  Interventions: Biological: Mycobacterium w; Other: Best standard care
- Best standard care (Active Comparator): Best standard care for sepsis
  Interventions: Other: Best standard care

INTERVENTIONS:
Biological: Mycobacterium w — Single daily dose of 0.3 mL of Mw (heat-inactivated Mw [0.5 × 10^9]; Immuvac, Cadila Pharma, Ahmedabad, India) in the deltoid region for 3 consecutive days
  Arms: Mycobacterium w group
Other: Best standard care — Antibiotics as early as possible; Norepinephrine > vasopressin > epinephrine for hypotension; Blood glucose 140-180 mg/dL; DVT and stress ulcer prophylaxis; Low tidal volume mechanical ventilation; Standard VAP, CLABSI prevention bundles

SUMMARY:
Recent evidence suggests that sepsis continuum includes an immune paralytic state, which may play a significant role in sepsis. Mycobacterium w by its TLR4 agonist activity may help in restoring immunity, thereby improving outcomes in patients with severe sepsis.

In this randomized trial, the investigators propose to evaluate the efficacy of Mw in patients with severe sepsis.

ELIGIBILITY:
Inclusion Criteria:

Patients with severe sepsis within 48 hours of first organ dysfunction

* Cardiovascular system dysfunction: systolic blood pressure ≤90 mm Hg or the mean arterial pressure ≤70 mm Hg for at least one hour despite adequate fluid resuscitation or the use of vasopressors to maintain a systolic blood pressure or mean arterial pressure of >90 and >65 mm Hg, respectively
* Renal dysfunction: urine output <0.5 ml/kg/hour for two consecutive hours despite adequate fluid resuscitation
* Respiratory system dysfunction: PaO2/FiO2 ≤300 or ≤250 if lung sepsis
* Hematologic dysfunction: platelet count <100,000/mm3 or decrease by 50% in the three days preceding enrollment
* Unexplained metabolic acidosis: pH ≤7.30

Exclusion Criteria:

* Pregnancy
* Gram-positive culture
* Only fungal infection as source of sepsis
* Patients who received cardiopulmonary resuscitation
* Those on immunosuppressive therapy
* Those unwilling to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Mortality | 28-day
  28-day all-cause mortality

SECONDARY OUTCOMES:
New onset organ dysfunction measured by delta SOFA (maximum minus baseline SOFA) | 28-day
  Measured by delta SOFA (maximum minus baseline SOFA)
Ventilator-free days | 28-day
  Day off the mechanical ventilator
Time-to-vasopressor withdrawal | 28-day
ICU length of stay | 28-day
Hospital length of stay | 28-day
New-onset infection | 28-day

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pulmonary Medicine, Chandigarh, Uttarakhand, India

REFERENCES:
- [Result] Sehgal IS, Agarwal R, Aggarwal AN, Jindal SK. A randomized trial of Mycobacterium w in severe sepsis. J Crit Care. 2015 Feb;30(1):85-9. doi: 10.1016/j.jcrc.2014.08.012. Epub 2014 Aug 28. PMID 25241089
- [Derived] Sehgal IS, Basumatary NM, Dhooria S, Prasad KT, Muthu V, Aggarwal AN, Pal A, Desai M, Chaudhry D, Supe PD, Kurmi P, Choudhuri R, Shah C, Agarwal R. A Randomized Trial of Mycobacterium w in Severe Presumed Gram-Negative Sepsis. Chest. 2021 Oct;160(4):1282-1291. doi: 10.1016/j.chest.2021.03.062. Epub 2021 May 7. PMID 33852919